CLINICAL TRIAL: NCT07187427
Title: Randomized Trial Comparing the Injection of Intrathecal Fentanyl Versus Epidural Fentanyl for the Initiation of Labour Analgesia on the Incidence of Pruritis.
Brief Title: Incidence of Pruritus Using Intrathecal Fentanyl Versus Epidural Fentanyl to Initiate Labour Analgesia.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Valerie Zaphiratos, Associate Professor of Anesthesiology, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2026-9304
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pruritis; Hypotension Drug-Induced; Urinary Retention; Fetal Bradycardia During Labor; Nausea and Vomitting; Satisfaction, Patient; Labor Analgesia; Neuraxial Opioid; Opioid Analgesic Adverse Reaction; Term Labour; Fentanyl Analgesia; Fentanyl Adverse Reaction
Keywords: neuraxial opioid induced pruritus during labor; Intrathecal fentanyl versus Epidural fentanyl
MeSH Terms: conditions — Pruritus; Hypotension; Urinary Retention; Nausea; Patient Satisfaction | interventions — Fentanyl; Analgesia, Epidural; Injections, Epidural

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups. The first group will receive an intrathecal injection of fentanyl, while the second will receive epidural fentanyl.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinal (Active Comparator): Intrathecal fentanyl This group will receive intrathecal Bupivacaïne 0.25% 1ml + Fentanyl 15mcg And epidural Nacl 0.9%
  Interventions: Procedure: Spinal analgesia
- Epidural (Active Comparator): Epidural fentanyl This group will receive intrathecal Bupivacaïne 0.25% 1ml + NaCl 0,9% And epidural fentanyl 100mcg
  Interventions: Procedure: Epidural Analgesia

INTERVENTIONS:
Procedure: Spinal analgesia — All procedures performed will be standardized. When neuraxial analgesia is required, an non-implicated anesthesiologist will performe the technique (not blind) The procedure will involve two steps. The first will involve an intraspinal injection of the solution using a 25-gauge Whitacre needle, while the second will be administered through the epidural catheter.
  STEP 1: Intraspinal SPINAL Group: Bupivacaine 0.25% Isobaric 1 ml + Fentanyl 15 mcg, (0,3ml)
  STEP 2: Epidural SPINAL group: 0.9% NaCl 2 ml.
  Other Names: Spinal; fentanyl
  Arms: Spinal
Procedure: Epidural Analgesia — All procedures performed will be standardized. When neuraxial analgesia is required, an non-implicated anesthesiologist will performe the technique (not blind) The procedure will involve two steps. The first will involve an intraspinal injection of the solution using a 25-gauge Whitacre needle, while the second will be administered through the epidural catheter.
  STEP 1: Intraspinal EPI Group: Bupivacaine 0.25% Isobaric 1 ml + NaCl 0.9% 0.3 ml
  STEP 2: Epidural EPI group: Fentanyl 100 mcg, (2 ml of a concentration of 50 mcg/ml)
  Other Names: Epidural; fentanyl
  Arms: Epidural

SUMMARY:
The purpose of this study is to investigate the effect of neuraxial analgesia initiation on the incidence of pruritus in laboring women. Specifically, this study aim to compare intrathecal fentanyl with epidural fentanyl in order to determine whether the epidural route is associated with a lower occurrence and severity of pruritus. By clarifying these differences, the research seek to optimize analgesic strategies during labor while minimizing opioid-related side effects

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Vaginal delivery
* Gestational age ≥ 37 weeks
* Requesting neuraxial analgesia
* French or English language

Exclusion Criteria:

* ASA score > 3
* Allergy or contraindication to receiving opioids/local anesthesia (morphine or fentanyl)
* BMI > 40 kg/m²
* Hepatic or renal failure,
* Severe preeclampsia and signs of severity according to the criteria of the American College of Obstetricians and Gynecologists
* Maternal hemorrhage (placental abruption, hepatic subcapsular hematoma,...)
* Severe scoliosis
* Biliary cholestasis or polymorphic eruption of pregnancy
* Inability to provide informed consent, either secondary to mental or physical disability or a significant language barrier (inability to understand English or French)
* Prior administration of an opioid or opioid misuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Pruritus | Every 15 minutes for the first hour, then every 30min for 2 hours until neuraxial analgesia
  Incidence et severity
  * 4-point Likert scale: Absent, light, moderate, severe/unbearable.
  * number of patients treated by antipruritic (Naloxone)

SECONDARY OUTCOMES:
Nausea Vomiting | 2 hours until neuraxial analgesia
  Incidence : Present or not Severity : number of patients treated (antinausea)
Hypotension | 2 hours until neuraxial analgesia
  Incidence : Decrease of arterial systolic pressure < 20% from basal Severity : Total dose of IV ephedrine
Urinary rentention | 24 hours until the neuraxial analgesia
  Number of urinary catheterizations
Maternal satisfaction | 24 hours until neuraxial analgesia
  Maternal satisfaction with neuraxial analgesia using :
  * Quality of Recovery-15 scale (QoR 15) : Score of 150 points to evaluate the recovery. The higher the score, the better the recovery.
  * Overall Benefit of Analgesia Score (OBAS) : multi-dimensional survey that assesses analgesia benefits, opioid-related adverse events, and patient satisfaction. Score of 28. The lowest the score, the better the benefits.
Fetal Bradycardia | 2 hours until neuraxial analgesia
  Incidence of fetal bradycardia Fetal monitoring is performed before and after the procedure. If a non-reassuring tracing is described by the obstetrical team, it will be noted in the patient's file. Fetal rhythm abnormalities via cardiotocogram are defined by nurses or obstetricians.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Sainte Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grangier L, Martinez de Tejada B, Savoldelli GL, Irion O, Haller G. Adverse side effects and route of administration of opioids in combined spinal-epidural analgesia for labour: a meta-analysis of randomised trials. Int J Obstet Anesth. 2020 Feb;41:83-103. doi: 10.1016/j.ijoa.2019.09.004. Epub 2019 Sep 23. PMID 31704251
- [Background] Kumar K, Singh SI. Neuraxial opioid-induced pruritus: An update. J Anaesthesiol Clin Pharmacol. 2013 Jul;29(3):303-7. doi: 10.4103/0970-9185.117045. PMID 24106351
- [Background] Wong CA, Scavone BM, Slavenas JP, Vidovich MI, Peaceman AM, Ganchiff JN, Strauss-Hoder T, McCarthy RJ. Efficacy and side effect profile of varying doses of intrathecal fentanyl added to bupivacaine for labor analgesia. Int J Obstet Anesth. 2004 Jan;13(1):19-24. doi: 10.1016/S0959-289X(03)00106-7. PMID 15321435
- [Background] Shah MK, Sia AT, Chong JL. The effect of the addition of ropivacaine or bupivacaine upon pruritus induced by intrathecal fentanyl in labour. Anaesthesia. 2000 Oct;55(10):1008-13. doi: 10.1046/j.1365-2044.2000.01618-2.x. PMID 11012498
- [Background] Palmer CM, Cork RC, Hays R, Van Maren G, Alves D. The dose-response relation of intrathecal fentanyl for labor analgesia. Anesthesiology. 1998 Feb;88(2):355-61. doi: 10.1097/00000542-199802000-00014. PMID 9477056
- [Background] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707